CLINICAL TRIAL: NCT01635868
Title: Long Term Recurrence and Chronic Pain After Repair for Small Umbilical or Epigastric Hernias. A Regional Cohort Study.
Brief Title: The Effect of Sutures Versus Mesh in Umbilical Hernia Repair
Acronym: ABSNOME
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume Christoffersen, MD, Hvidovre University Hospital
Other Study IDs: ABSNOME
Record Dates: First submitted 2012-07-04; First posted 2012-07-10 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Ventral Hernia Midline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- umbilical hernia repair: patients having umbilical or epigastric hernia repair from 2008-2010 in Zealand

SUMMARY:
Background Mesh repair reduces the risk of reoperation for recurrence in patients with small umbilical and epigastric hernias compared with sutured repair. However, reoperation for recurrence underestimates total recurrence (reoperation or clinical) and mesh reinforcement may induce chronic pain. This study investigated the cumulated risk of recurrence after open mesh and sutured repair in small (≤2 cm) umbilical and epigastric hernias. Possible risk factors were evaluated for chronic pain and recurrence.

Methods A cohort study with questionnaire-follow-up was conducted. Patients with primary, elective, open mesh or sutured repair for a small umbilical or epigastric hernia (≤2 cm) were included. Follow-up was performed by a validated questionnaire regarding suspicion of recurrence and chronic pain (moderate or severe). Suspected recurrence qualified for clinical examination. Recurrence was defined as reoperation for recurrence or clinical recurrence. Risk factors for recurrence and chronic pain were investigated by multivariate analyses.

Results

1 313 patients completed the questionnaire and/or clinical follow-up (83 % response rate) and follow-up time was median 40 months (range 0-66 months). The total cumulated recurrence rate 55 months after primary repair was 10 % for mesh repair and 21 % for sutured repair (P=0.001). The incidence of chronic pain was 6 % after mesh repair and 5 % after sutured repair (P = 0.711). Recurrence was the only independent risk factor for chronic pain (P<0.001).

Conclusion Mesh repair halved the long-term risk of recurrence after repair for small umbilical and epigastric hernias without increased risk of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* elective open mesh or sutured repair of small umbilical or epigastric hernia repairs

Exclusion Criteria:

* acute operation
* operation outside region of Zealand
* laparoscopic repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient having mesh or sutured repair of small (> 2 cm) umbilical or epigastric hernias in the region of Zealand from 1th of January 2008 to 31th of December 2010.
Sampling Method: Non-Probability Sample
Enrollment: 1313 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
recurrence (clinical or reoperation for recurrence) | 3 years
  follow-up time will be from 3-5 years

SECONDARY OUTCOMES:
chronic pain | 3-5 years after surgery
  patient self-registration on VRS. Moderate or severe pain is regarded as chronic pain

OTHER OUTCOMES:
risk factors for recurrence and chronic pain | 3-5 yrs
  We identify risk factor for chronic pain and recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bisgaard, DMSc, Study Director — University Hospital of Copenhagen Hvidovre
Locations (1):
- Hvidovre Hospital University of Copenhagen, Hvidovre, Denmark